CLINICAL TRIAL: NCT06586242
Title: A Two Arm, Randomized, Prospective, Multicenter Study of Penpulimab Combined With Anlotinib Hydrochloride and Chemotherapy in the Perioperative Treatment of Locally Advanced Resectable Esophageal Cancer
Brief Title: Efficacy and Safety of Penpulimab Combined With Anlotinib and Chemotherapy
Acronym: EASOPCWAAC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TQXB-E-002
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- penpulimab combined with anlotinib hydrochloride plus albumin paclitaxel and oxaliplatin (Experimental): penpulimab：200mg, intravenous infusion, 30-60 minutes per infusion, once every 3 weeks, administered on the first day of each cycle anlotinib hydrochloride：Body weight <60kg, 8mg Po, body weight ≥ 60kg, 10mg Po, D 1-14, q3w Albumin paclitaxel: 260mg/m2, intravenous infusion, 30 minutes per infusion, once every 3 weeks, d 1 medication per week oxaliplatin：130mg/m2, i.v., administered after albumin paclitaxel, on day 1 of each week; Three weeks is a treatment cycle.
  Interventions: Drug: Penpulimab;Anlotinib;albumin paclitaxel;oxaliplatin;lobaplatin
- penpulimab combined with anlotinib hydrochloride plus albumin paclitaxel and lobaplatin (Active Comparator): penpulimab：200mg, intravenous infusion, 30-60 minutes per infusion, once every 3 weeks, administered on the first day of each cycle anlotinib hydrochloride：Body weight <60kg, 8mg Po, body weight ≥ 60kg, 10mg Po, D 1-14, q3w Albumin paclitaxel: 260mg/m2, intravenous infusion, 30 minutes per infusion, once every 3 weeks, d 1 medication per week lobaplatin：50mg/m2, i.v., administered after albumin paclitaxel, on day 1 of each week; Three weeks is a treatment cycle.
  Interventions: Drug: Penpulimab;Anlotinib;albumin paclitaxel;oxaliplatin;lobaplatin

INTERVENTIONS:
Drug: Penpulimab;Anlotinib;albumin paclitaxel;oxaliplatin;lobaplatin — 200mg, intravenous infusion, 30-60 minutes per infusion, once every 3 weeks, Penpulimab:administered on the first day of each cycle Anlotinib:Body weight <60kg, 8mg Po, body weight ≥ 60kg, 10mg Po, D 1-14, q3w
  Other Names: AK105；AL3818

SUMMARY:
This study is a two arm, randomized, prospective, multicenter study on the perioperative treatment of locally advanced resectable esophageal cancer with penpulimab combined with anlotinib hydrochloride and chemotherapy.

DETAILED DESCRIPTION:
The study was a two arm, randomized, prospective, multicenter study. The experimental group was treated with penpulimab combined with anlotinib hydrochloride plus albumin paclitaxel and oxaliplatin, and the control group was treated with penpulimab combined with anlotinib hydrochloride plus albumin paclitaxel and lobaplatin

ELIGIBILITY:
Inclusion Criteria:

* 1. only those who meet all the following requirements can be enrolled in this trial: 1. age 18-75 years old, both male and female;
* 2. according to gastroscope / ultrasonic gastroscope biopsy, the pathology suggests esophageal cancer, and the clinical diagnosis is ct2n1-3m0 or ct3n0-3m0 or ct4n0-3m0, and the TNM stage is stage ii-iva;
* 3. patients with non cervical esophageal cancer;
* 4. have not received previous systemic and local treatment for esophageal cancer according to RECIST 1 1 criteria at least one measurable lesion was used for imaging evaluation of neoadjuvant therapy;
* 5.ecog PS: 0-1 point;
* 6. estimated survival ≥ 12 months;
* 7. the subject had no dysfunction of major organs, and the investigator assessed that the thyroid, lung, bone marrow, liver, kidney and heart functions were basically normal; 8. women of childbearing age must have taken reliable contraceptive measures or had a pregnancy test (serum or urine) within 7 days before enrollment, and the results are negative, and are willing to use appropriate methods of contraception during the test and - 8 weeks after the last administration of test drugs. For men, they must agree to use appropriate methods of contraception or have been surgically sterilized during the trial and 8 weeks after the last administration of the trial drug;
* 9. the subjects voluntarily joined the study, signed the informed consent, had good compliance, followed the planned schedule, actively cooperated with returning to the hospital for regular clinical follow-up and necessary treatment, and cooperated with regular blood and tissue sample acquisition.

Exclusion Criteria:

* 1. 5 years of other malignant tumors, except for cured cervical carcinoma in situ, non melanoma skin cancer and superficial bladder tumor [ta (non invasive tumor), tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)];
* 2. patients with ulcerative esophageal squamous cell carcinoma;
* 3. patients with esophageal fistula or tracheal fistula;
* 4. those who are sensitive to anlotinib, pembrolizumab, albumin paclitaxel or oxaliplatin and excipients;
* 5. have a history of immune deficiency, including HIV positive or suffering from other acquired or congenital immune deficiency diseases, or have a history of organ transplantation;
* 6. patients with any severe and / or uncontrolled disease, including:

  1) Patients with unsatisfactory blood pressure control (systolic blood pressure ≥ 160 mm Hg or diastolic blood pressure ≥ 100 mmHg); 2) Myocardial ischemia or myocardial infarction of grade I or above; 3) Arrhythmia (including QT interval ≥ 480 MS) and grade I cardiac insufficiency; 4) Diabetes mellitus with poor blood glucose control (fasting blood glucose (FBG) >10mmol/l) or high-dose glucocorticoid treatment; 5) Active or uncontrolled severe infection; 6) Decompensated liver disease, active hepatitis B (HBV-DNA ≥ 104copies/ml or 2000iu/ml) or hepatitis C (hepatitis C antibody and HCV RNA positive) were all above the lower limit of the analysis method; 7) Hyperthyroidism and hypothyroidism; 8) Active tuberculosis.
* 7. unrelieved toxic reactions higher than CTCAE grade 1 due to any previous treatment, excluding hair loss;
* 8. esophageal cancer patients with active bleeding within 2 months of the primary lesion;
* 9. patients whose tumors have invaded the important blood vessels or are judged by the investigator to be very likely to invade the important blood vessels during the follow-up study and cause fatal massive hemorrhage;
* 10. patients with multiple factors affecting oral drugs (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.), but patients with dysphagia who can drink water, can take anlotinib after dissolving the particles;
* 11. the urine routine indicates that the urine protein is ≥ + +, and the 24-hour urine protein quantitation is confirmed to be >1.0 g;
* 12. received major surgical treatment, incision biopsy or obvious traumatic injury within 28 days before grouping;
* 13. abnormal coagulation function: inr>1.5 or prothrombin time (PT) >uln+4 seconds or APTT >1.5uln), with bleeding tendency or undergoing thrombolytic or anticoagulant therapy; Within 4 weeks before grouping, patients with any bleeding or bleeding events ≥ CTCAE grade 3 had unhealed wounds, ulcers or fractures;
* 14. Those who have had arterial / venous thrombotic events within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism;
* 15. pregnant or lactating women;
* 16. patients with distant metastasis;
* 17. patients with significant myelosuppression;
* 18. have a history of mental illness or abuse of psychotropic drugs;
* 19. Patients who have participated in clinical trials of other drugs within 4 weeks;
* 20. according to the judgment of the investigator, patients with concomitant diseases that seriously endanger the safety of patients or affect the completion of the study;
* 21. the investigator believes that it is not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2036-04 (Estimated)

PRIMARY OUTCOMES:
the Pathological complete response (PCR) rate | 2years
  Pathological complete response (PCR) rate

SECONDARY OUTCOMES:
the rate of R0 resection | 2years
  R0 resection rate
Disease free survival time | 2years
  Disease free survival
1-year OS rate | 2years
  1-year OS rate

CONTACTS AND LOCATIONS:
Overall Officials: Liu Hong, Master, Principal Investigator — The First Affiliated Hospital of Air Force Medical University
Locations (1):
- The First Affiliated Hospital of the Air Force Medical University, Xi'an, Shaan'xi, China